CLINICAL TRIAL: NCT06472024
Title: Effects Of Manual Acupuncture On Mucositis Due To Radiotherapy For Nasopharynx Cancer On Visual Analogue Scale (Vas) Score And Quality Of Life
Brief Title: Assessing Manual Acupuncture's Impact on Mucositis From Nasopharynx Cancer Radiotherapy: A Visual Analogue Scale (VAS) and Quality of Life Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Imelda Dimara, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-05-0717
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Nasopharyngeal Carcinoma; Mucositis
MeSH Terms: conditions — Neoplasms; Nasopharyngeal Carcinoma; Mucositis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Acupuncture (Experimental): The verum acupuncture group will receive actual acupuncture therapy 2 times per week for 3 weeks
  Interventions: Procedure: Verum Acupuncture
- Sham Acupuncture (Sham Comparator): The Sham acupuncture group will receive Sham acupuncture therapy 2 times per week for 3 weeks
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Verum Acupuncture — Acupuncture therapy uses filiform needles at a perpendicular angle at acupuncture points to produce a therapeutic effect.
  Arms: Verum Acupuncture
Procedure: Sham Acupuncture — Sham Acupuncture therapy uses filiform needles but is only attached with tape to acupuncture points
  Arms: Sham Acupuncture

SUMMARY:
The goal of this clinical trial is to learn if acupuncture can play a role in reducing pain and improving the quality of life of post-radiotherapy nasopharyngeal cancer mucositis patients. The main questions it aims to answer are:

- Do manual acupuncture and medication therapy affect pain intensity as measured by the visual analogue scale (VAS) in patients with oral mucositis compared with sham manual acupuncture and medication?

Participants will receive acupuncture therapy 2 times a week for 3 weeks

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate the role of acupuncture in pain relief and improving the quality of life of nasopharyngeal cancer patients with post-radiotherapy mucositis. Participants were 30 men/females with mucositis in post-radiotherapy nasopharyngeal cancer aged 19-59 years. They will be divided into 2 groups: (1) verum acupuncture and (2) sham acupuncture. Acupuncture is scheduled 2 times per week for 3 weeks. Research assessment on pain scale and improvement in quality of life

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been proven by anatomical pathology examination to have a diagnosis of Nasopharyngeal Cancer.
* Subjects with adult Nasopharyngeal Cancer aged 19 years - 59 years.
* Nasopharyngeal Cancer Patients, who underwent bilateral Head and Neck radiotherapy.
* Patients diagnosed with mucositis.
* Willing to participate in the research until completion by signing an informed consent.

Exclusion Criteria:

* Nasopharyngeal Cancer patients who have distant metastases (based on the Tumor Node Metastasis (TNM) classification with the presence of metastases (M1)).
* Subjects who still smoke and consume alcohol to date.
* Patients have contraindications for manual acupuncture, namely the use of anti-coagulant drugs, the presence of infection or wounds at the puncture site, emergency conditions, and pregnancy.
* There is a history of allergy to stainless steel materials.
* Patients with blood clotting disorders; Platelets <50,000/μL, Absolute Neutrophil Count (ANC) <1000/mm3, patients undergoing anticoagulant therapy with International Normalized Ratio (INR) >2.47

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Monitored 2 times per week for 3 weeks, and followed up again at week 4 without intervention.
  VAS is used to assess pain complaints on a scale of 1-10. The VAS scale consists of: mild pain scale 1-3, moderate pain scale 4-6 and severe pain scale 7-10
European Organization For Research And Treatment Of Cancer Head and Neck Cancer Quality of Life Questionnaire (EORTC QLQ-H&N35) | Monitored before and after intervention. After the intervention; Results will be measured at week 3 after intervention and results will be measured at week 4 without intervention.
  The EORTC QLQ-H&N35 is a questionnaire designed to assess the health-related quality of life in patients with head and neck cancer. It consists of 35 questions covering various aspects such as pain, swallowing, speech, social eating, and emotional functioning. Each question is scored on a scale from 1 to 4, with 1 representing "not at all" and 4 representing "very much".
  To calculate a score for each domain, the individual item scores are averaged. Higher scores indicate more severe symptoms or poorer quality of life in that domain. Additionally, there are specific guidelines provided by the European Organization for Research and Treatment of Cancer (EORTC) for scoring and interpreting the results, with a minimum and maximum scale of 0-33: mild, 34-66: moderate, 67-100: severe.

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - RSCM

IPD SHARING:
Plan to Share IPD: No